CLINICAL TRIAL: NCT06309901
Title: Comparison of Facial Distortion Model and Instrument Assisted Soft Tissue Mobilization (IASTM) Techniques After Arthroscopic Meniscus Repair
Brief Title: Facial Distortion Model and Instrument Assisted Soft Tissue Mobilization Techniques
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Bahar Anaforoglu Külünkoglu, Assoc. Prof., Ankara Yildirim Beyazıt University
Other Study IDs: ankaraYBU2019-199
Record Dates: First submitted 2024-02-16; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Meniscus Injury
Keywords: IASTM; FDM; Meniscus repair
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group: A progressive home exercise program consisting of 3 phases was applied.
  Interventions: Other: Exercise
- FDM Group: In addition to the progressive home exercise program consisting of 3 phases, the trigger band technique of the fascial distortion model was applied around the knee.
  Interventions: Other: Exercise; Other: Fascial Distortion Model
- IASTM Group: In addition to the progressive home exercise program consisting of 3 phases, the IASTM was applied with Graston technique around the knee.
  Interventions: Other: Exercise; Other: Instrument Assisted Soft Tissue Mobilisation

INTERVENTIONS:
Other: Exercise — Home exercises were applied in 3 progressive phases.
  1st phase: postoperative 0-4. week, 2nd phase: 5-12. week, 3rd phase 12-15. week.
  In the 1st phase, ice application, strengthening for the hip, knee and ankle, and walking exercises were applied. 90 degrees knee flexion range of movement (ROM) was targeted.
  In the 2nd phase, the resistance of the strengthening exercises was increased and closed kinetic chain exercises were added. Weight bearing, step climbing and balance exercises were performed. Full ROM targeted in the knee.
  In the 3rd phase, pain-free full ROM was targeted, and progressive strengthening, balance and agility exercises for sports and recreational activities were applied.
Other: Fascial Distortion Model — At the beginning of the 2nd phase of the treatment, starting from the 5th week, twice a week for 4 weeks, a total of 8 sessions of FDM technique were applied.
  In this study, trigger band technique was chosen to apply around the knee. Interventions were made directly to the skin in the form of medial, lateral, anterior, posterior techniques of the knee and posterior and lateral techniques of the thigh. The techniques was made after the exercises.
  Groups: FDM Group
Other: Instrument Assisted Soft Tissue Mobilisation — At the beginning of the 2nd phase of the treatment, starting from the 5th week, twice a week for 4 weeks, a total of 8 sessions of IASTM technique were applied.
  In this study, the Graston technique was chosen to apply IASTM around the knee. Technique was applied with using stainless steel and ultrasound gel to around the knee, m. quadriceps, m. hamstring, iliotibial band and medial thigh. The technique was performed for at least 2 minutes in each region.
  Groups: IASTM Group

SUMMARY:
To compare the effects of facial distortion model and equipment assisted soft tissue mobilization techniques on the treatment process, which are among the applications in the rehabilitation process after meniscus repair.

DETAILED DESCRIPTION:
It is possible that pain, ROM, lower extremity flexibility and knee functions will be negatively affected after arthroscopic meniscus repair. This study searches and compares the effectiveness of fascial distortion model (FDM) and IASTM methods for these parameters that can be affected.

ELIGIBILITY:
Inclusion Criteria:

* The meniscus rupture and suspected magnetic resonance (MR) were diagnosed and operated by the surgeon during arthroscopy.
* Those treated with the same surgical technique
* Can walk independently before the operation
* Can continue treatment for 4 weeks
* Without chondral damage
* Can continue treatment for 4 weeks
* Those who have not had lower extremity surgery before
* No fracture to prevent load transfer in the last 6 months
* There is no full rupture of any ligament in the knee
* Without knee instability
* Those without abnormal changes in Q angle
* According to Cooper classification, meniscus affected area is not in A and F regions.
* Without protruded or extruded herniated disc
* There is no contract in the directory

Exclusion Criteria:

* Can not continue treatment for 4 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals who were diagnosed after meniscus tear between 18-55 years and suspected magnetic resonance (MRI) or operated during arthroscopy and operated by the surgeon, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Change from postoperative 4. week at 8. week
  It is used to convert some values that cannot be measured numerically into numerical values. Two end definitions of the parameter to be evaluated on both ends of a 100 mm line are written and the patient is asked to indicate where his / her condition is appropriate on this line by drawing a line or by marking or pointing.
environmental measurement | Change from postoperative 4. week at 8. week
  One of the anthropometric measurement techniques is measured using tape measure. Medial tibial plateau and 5 cm intervals at 5 cm, 10 cm and 15 cm points are marked and the circumference of the knee and the leg is measured.
Power Track Manuel Muscle Tester | Change from postoperative 4. week at 8. week
  In the manual muscle test, a hand dynamometer was developed for the standardization of the given resistance, which determines the resistance given by the tester. This tool objectively shows the amount of force used in muscle testing. The tool is placed proximal to the tibia, the amount of force applied is read from the manometer on the dorsal side of the hand. It is placed on the front for extension and on the back for flexion.
sit and reach test | Change from postoperative 4. week at 8. week
  To reach the farthest in a sitting position.
Goniometric measurement | Change from postoperative 4. week at 8. week
  uses a goniometer to measure the hamstring flexibility during a passive straight leg lift.
The Western Ontario Meniscal Evaluation Tool (WOMET ) | Change from postoperative 4. week at 8. week
  In this inventory, there are 16 items that represent physical domains (nine items), sports / entertainment / work / lifestyle (four items) and the domains of emotions (three items). A value between 0-10 is requested in each item. The score of each subgroup is obtained by dividing the marked values of the questions of that section by the number of questions and multiplying by 10. The total score is obtained by summing all scores and dividing by 16 and multiplying by 10.
Lysholm Knee Score | Change from postoperative 4. week at 8. week
  It is a scoring questioning situations such as pain, stair climbing, squatting, walking pattern and swelling of the knee while showing certain activities. In the Lysholm scoring system; It can be classified as 0-20 bad, 21-40 medium, 41-60 medium-good, 61-80 good, 81-100 perfect.

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Anaforoğlu, Assoc. Prof., Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Yıldırım Beyazıt University Yenimahalle Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
has not been decided yet.

REFERENCES:
- [Result] Cheatham SW, Lee M, Cain M, Baker R. The efficacy of instrument assisted soft tissue mobilization: a systematic review. J Can Chiropr Assoc. 2016 Sep;60(3):200-211. PMID 27713575
- [Result] Kalichman L, Ben David C. Effect of self-myofascial release on myofascial pain, muscle flexibility, and strength: A narrative review. J Bodyw Mov Ther. 2017 Apr;21(2):446-451. doi: 10.1016/j.jbmt.2016.11.006. Epub 2016 Nov 14. PMID 28532889
- [Result] Thalhamer C. A fundamental critique of the fascial distortion model and its application in clinical practice. J Bodyw Mov Ther. 2018 Jan;22(1):112-117. doi: 10.1016/j.jbmt.2017.07.009. Epub 2017 Jul 25. PMID 29332733